CLINICAL TRIAL: NCT03898102
Title: Zinc Supplement in Metastatic Colorectal Cancer Patients Receiving Regorafenib: Phase II Prospective Randomized Trial
Brief Title: Zinc Supplement in Regorafenib Treated mCRC Patient
Acronym: ZnCORRECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yeh Chun-Nan, Professor and Director, Division of General Surgery, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1901090003
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regorafenib treatment with Zn supplement (Experimental): Patients enrolled in this arm received regorafenib with zinc supplementation to examine if zinc supplementation can decrease the incidence of grade 2 or higher HFSR.
  Interventions: Drug: Regorafenib; Dietary Supplement: Zinc gluconate supplement
- Regorafenib treatment only (Active Comparator): Patients enrolled in this arm received regorafenib without zinc supplementation, which is the standard treatment of patients of metastatic colorectal cancer who failed previous standard therapy.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — regorafenib plus zinc gluconate
Dietary Supplement: Zinc gluconate supplement — Zinc gluconate supplement
  Arms: Regorafenib treatment with Zn supplement

SUMMARY:
Phase II randomized trial to investigate whether supplementation of zinc decreases the incidence of HFSR that occurs after treatment of tyrosine kinase inhibitor, regorafenib.

DETAILED DESCRIPTION:
This study is aimed to investigate the effect of zinc supplementation on improving regorafenib treatment safety and efficacy in patients with metastatic colorectal cancer (mCRC). The difference in grade 2 or worse hand-foot skin reaction (HFSR) incidence within the first 8 weeks of regorafenib treatment between two arms will be examined as the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mCRC who have been previously treated with, or are not considered candidates for, other locally approved standard treatment(s) and for whom the decision has been made per investigator's routine treatment practice to prescribe regorafenib
* Ability to understand and willingness to sign written Informed Consent Form (ICF)

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice
* Patients with baseline Zinc level above 120 ug/dL
* Patients with known allergy to Zinc supplementation
* Pregnancy
* Patients who are unsuitable for study participation, based on investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Difference in grade 2 or worse HFSR incidence within the first 8 weeks of regorafenib treatment between mCRC patients who receive regorafenib treatment with or without zinc supplementation | 8 weeks
  Percentages

SECONDARY OUTCOMES:
Percentage of zinc deficiency before and after regorafenib treatment at weeks 4 | 4 weeks
  Percentages
Percentage of zinc deficiency before and after regorafenib treatment at weeks 8 | 8 weeks
  Percentages
Percentage of regorafenib dose reduction | Through study completion, estimated 2 years
  Percentages
Progression Free Survival (PFS) | Through study completion, estimated 2 years
  months
Objective tumor response rate (ORR) | Through study completion, estimated 2 years
  rate
Disease control rate (DCR) | Through study completion, estimated 2 years
  rate
Overall survival (OS) | Through study completion, estimated 2 years
  months
Duration of treatment of regorafenib (DoT) | through study completion, estimated 2 years
  months

OTHER OUTCOMES:
Percentage of patients with clinically significant finding in physical examination results, as assessed by general appearance | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically significant finding in physical examination results, as assessed by HEENT (head, eyes, ears, nose, and throat) | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically significant finding in physical examination results, as assessed by mouth | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically significant finding in physical examination results, as assessed by skin | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically significant finding in physical examination results, as assessed by neck (thyroid gland included) | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically significant finding in physical examination results, as assessed by lymph nodes | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically important change in vital sign results from baseline, as assessed by systolic pressure | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically important change in vital sign results from baseline, as assessed by diastolic blood pressure | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically important change in vital sign results from baseline, as assessed by pulse rate | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically important change in vital sign results from baseline, as assessed by respiratory rate | Through study completion, estimated 2 years
  Percentage
Percentage of patients with clinically important change in vital sign results from baseline, as assessed by body temperature | Through study completion, estimated 2 years
  Percentage
Percentage of patients with significant changes from baseline in clinical laboratory test results, assessed by hematology panel | Through study completion, estimated 2 years
  Percentage
Percentage of patients with significant changes from baseline in clinical laboratory test results, assessed by biochemistry panel | Through study completion, estimated 2 years
  Percentage
Percentage of patients with adverse events (graded by NCI-CTCAE v4.03) | Through study completion, estimated 2 years
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Nan Yeh, MD, Principal Investigator — Chang Gung Memorial Hospital

REFERENCES:
- [Derived] Huang WK, Hsu HC, Yang TS, Lu CW, Pan YR, Wu CE, Chung WH, Hung SI, Yeh CN. Zinc supplementation decreased incidence of grade >/=2 hand-foot skin reaction induced by regorafenib: A phase II randomized clinical trial. Eur J Cancer. 2023 Dec;195:113286. doi: 10.1016/j.ejca.2023.113286. Epub 2023 Nov 13. PMID 37968194